CLINICAL TRIAL: NCT00943059
Title: The Effect of Lipid Lowering by Acipimox on Cardiac and Skeletal Muscle Mitochondrial Function
Brief Title: Cross-over Study on Effect of Lipid Lowering by Acipimox on Cardiac and Skeletal Muscle Mitochondrial Function
Acronym: ACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Center for Translational Molecular Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 09-3-033; CTMM2008172; EFSD10122008; ZonMw91896618
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 2; Cardiomyopathy, Dilated
Keywords: Mitochondrial function; Diabetes; Cardiomyopathy; insulin resistance; lipid lowering; triglycerides; Acipimox
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiomyopathy, Dilated; Diabetes Mellitus; Cardiomyopathies; Insulin Resistance | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acipimox (Experimental): Subjects will receive Acipimox or a placebo in random order. Acipimox is a commercially available and registrated drug, that lowers free fatty acids by inhibiting hormone sensitive lipase in the peripheral adipose tissue. No serious side-effects are known other than rare anaphylactic reactions.
  Interventions: Drug: Acipimox
- Cellulosum mycrocryst capsula (Placebo Comparator): Subjects will receive Acipimox or a placebo in random order. Acipimox is a commercially available and registrated drug, that lowers free fatty acids by inhibiting hormone sensitive lipase in the peripheral adipose tissue. No serious side-effects are known other than rare anaphylactic reactions.
  Interventions: Drug: Cellulosum Mycrocryst

INTERVENTIONS:
Drug: Acipimox — A capsula is given with 250mg Acipimox, 3dd; 1 after each meal. This will be done during 14 days.
  Other Names: Olbetam; Nedios
  Arms: Acipimox
Drug: Cellulosum Mycrocryst — Capsule with cellulosum powder; this has to be taken 3 dd; 1 after each meal during 14 days.
  Other Names: Placebo
  Arms: Cellulosum mycrocryst capsula

SUMMARY:
Accumulation of lipid in skeletal and cardiac muscle has been associated with insulin resistance and diabetic cardiomyopathy. In skeletal muscle, lipotoxic damage has been suggested to lead to dysfunction of mitochondria. It remains unknown whether lipotoxicity leads to mitochondrial dysfunction in heart as well, and if so, whether this also leads to cardiomyopathy (failure of the heart). Although it has been shown that lipid lowering agents can improve insulin sensitivity, the effect of lowering free fatty acids on cardiac and skeletal muscle mitochondrial function remains unknown. In this study the investigators want to investigate whether lowering cardiac and muscular lipid content will improve mitochondrial and cellular function in type 2 diabetic patients.

To this end, type 2 diabetic patients and body mass index (BMI)-matched controls will be included in a blinded cross-over design, in which subjects will receive a lipid lowering agent (Acipimox) or placebo for 2 weeks in random order. During treatment, diabetes medication will be stopped. Baseline measurements will be performed prior to the study and after each treatment to assess cardiac and muscular lipid accumulation, cardiac function, mitochondrial function and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal females
* Age 40-70 years
* Obese (BMI > 30 kg/m2), non-insulin dependent type 2 diabetic patients and BMI matched control subjects without diabetes.
* Generally healthy with specifically no known cardiovascular disease, dyslipidemia, or gastric ulcers (contra-ind. of Acipimox), which can affect the study parameters.
* Must be on sulphonylurea(SU)- derivate or metformin therapy for at least six months with a constant dose for at least two months, or on dietary treatment for at least six months
* Well-controlled diabetes: HbA1c<8%.
* Control subjects must have a plasma glucose lower than 6,1 mmol/L.
* Stable dietary habits (no weight loss/gain > 3 kg in the last 6 months)

Exclusion Criteria:

* Known cardiovascular disease, dyslipidemia, hepatic or renal failure and gastric ulcers.
* Insulin dependent Diabetic patients.
* Use of lipid lowering agents, except from Statins, as these do not affect triglycerides levels (with exception to Lipitor).
* Use of Thiazolidines (glitazone/rosiglitazone/pioglitazone/troglitazone)
* Use of anti-coagulants (not thrombocyte-aggregation inhibitors)
* Aberrant ECG (with signs of ischemia or cardiac failure or arrythmia's)
* Weight gain/loss > 3 kg in the last 6 months.
* Hb < 7,3 in women, and < 7,8 in men.
* Contraindications for MRI scans:

  * Electronic implants such as pacemakers or neurostimulator
  * Iron-containing corpora aliena in eyes or brain
  * Some hearing aids and artificial (heart) valves which are contraindicated for MRS
  * Claustrophobia
* Subjects, who do not want to be informed about unexpected medical findings, or do not wish that their physician is informed, cannot participate in the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
changes in mitochondrial function | 2 weeks
changes in cardiac function | 2 weeks
lipid accumulation in ectopic tissue (cardiac and skeletal muscle) | 2 weeks

SECONDARY OUTCOMES:
insulin sensitivity | 2 weeks
oxidative stress markers | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Background] Schrauwen-Hinderling VB, Kooi ME, Hesselink MK, Jeneson JA, Backes WH, van Echteld CJ, van Engelshoven JM, Mensink M, Schrauwen P. Impaired in vivo mitochondrial function but similar intramyocellular lipid content in patients with type 2 diabetes mellitus and BMI-matched control subjects. Diabetologia. 2007 Jan;50(1):113-20. doi: 10.1007/s00125-006-0475-1. Epub 2006 Nov 9. PMID 17093944
- [Background] Phielix E, Schrauwen-Hinderling VB, Mensink M, Lenaers E, Meex R, Hoeks J, Kooi ME, Moonen-Kornips E, Sels JP, Hesselink MK, Schrauwen P. Lower intrinsic ADP-stimulated mitochondrial respiration underlies in vivo mitochondrial dysfunction in muscle of male type 2 diabetic patients. Diabetes. 2008 Nov;57(11):2943-9. doi: 10.2337/db08-0391. Epub 2008 Aug 4. PMID 18678616
- [Background] De Feyter HM, Lenaers E, Houten SM, Schrauwen P, Hesselink MK, Wanders RJ, Nicolay K, Prompers JJ. Increased intramyocellular lipid content but normal skeletal muscle mitochondrial oxidative capacity throughout the pathogenesis of type 2 diabetes. FASEB J. 2008 Nov;22(11):3947-55. doi: 10.1096/fj.08-112318. Epub 2008 Jul 24. PMID 18653763
- [Background] Schrauwen-Hinderling VB, Roden M, Kooi ME, Hesselink MK, Schrauwen P. Muscular mitochondrial dysfunction and type 2 diabetes mellitus. Curr Opin Clin Nutr Metab Care. 2007 Nov;10(6):698-703. doi: 10.1097/MCO.0b013e3282f0eca9. PMID 18089950
- [Derived] Houzelle A, Jorgensen JA, Schaart G, Daemen S, van Polanen N, Fealy CE, Hesselink MKC, Schrauwen P, Hoeks J. Human skeletal muscle mitochondrial dynamics in relation to oxidative capacity and insulin sensitivity. Diabetologia. 2021 Feb;64(2):424-436. doi: 10.1007/s00125-020-05335-w. Epub 2020 Nov 30. PMID 33258025
- [Derived] Phielix E, Jelenik T, Nowotny P, Szendroedi J, Roden M. Reduction of non-esterified fatty acids improves insulin sensitivity and lowers oxidative stress, but fails to restore oxidative capacity in type 2 diabetes: a randomised clinical trial. Diabetologia. 2014 Mar;57(3):572-81. doi: 10.1007/s00125-013-3127-2. Epub 2013 Dec 6. PMID 24310562
- See also: Website of location of trail. — http://www.maastrichtuniversity.nl
- See also: Website of department of Human Biology, who conduct trail. — http://www.hb.unimaas.nl/